CLINICAL TRIAL: NCT00004643
Title: Phase II Pilot Study of Cytarabine for Refractory Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Michigan (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 199/11685; UMMC-91208
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-03

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: arthritis & connective tissue diseases; immunologic disorders and infectious disorders; rare disease; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis; Connective Tissue Diseases; Immune System Diseases; Communicable Diseases; Rare Diseases | interventions — Cytarabine

INTERVENTIONS:
Drug: cytarabine

SUMMARY:
OBJECTIVES: I. Evaluate the toxicity of cytarabine in patients with refractory systemic lupus erythematosus.

II. Evaluate objective disease parameters, including serum complement levels, anti-DNA antibody titers, sedimentation rate, and the systemic lupus activity measure in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Subcutaneous cytarabine is given for 5 days. Patients are re-treated every 4 weeks for a maximum of 3 courses; those who relapse prior to the second course are re-treated every 3 weeks.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Disease Characteristics

* Clinically documented active systemic lupus erythematosus demonstrating at least 4 revised diagnostic criteria
* Unresponsive to conventional therapy with nonsteroidal anti-inflammatory drugs (NSAIDs), topical corticosteroids, and antimalarials
* Intolerable side effects from corticosteroids or other immunosuppressive drugs Failure on immunosuppressives not required
* No life-threatening disease, e.g.: Lupus cerebritis Rapidly progressive glomerulonephritis

Prior/Concurrent Therapy

* No concurrent other DNA synthesis inhibitors, NSAIDs, and prednisone continued on study

Patient Characteristics

* Hematopoietic: WBC at least 2000; Platelets at least 100,000
* Renal: Creatinine clearance at least 20 mL/min
* Other: No major infection within 2 weeks prior to entry
* Negative pregnancy test required of fertile women
* Effective contraception required of fertile women. Advised for men during and for 75 days after therapy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10
Dates: Start 1995-02

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Richardson, Study Chair — University of Michigan

REFERENCES:
- [Background] Yung RL, Richardson BC. Cytarabine therapy for refractory cutaneous lupus. Arthritis Rheum. 1995 Sep;38(9):1341-3. doi: 10.1002/art.1780380926. No abstract available. PMID 7575733